CLINICAL TRIAL: NCT07202325
Title: A Self-Help Intervention to Improve Functioning, Symptoms, and Treatment Utilization Among Non-Treatment Engaged Post 9/11 Veterans With Depression or PTSD Symptoms
Brief Title: Self-Help Intervention for Post 9/11 Veterans With Depression or PTSD Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRD4-013-24W; RD000544 (Other Grant/Funding Number: VA Brain, Behavioral and Mental Health)
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Depression; Stress Disorders, Post-Traumatic
Keywords: Self-Management; Depression; Post Traumatic Stress Disorder; Veterans; Psychosocial Functioning; Clinical Trial; Psychological Intervention; Self-Help
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial in which participants are randomized to either the intervention condition (REST-V) or control (standard resources) condition.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention condition (Experimental): Self-help intervention
  Interventions: Behavioral: Resilience Training for Veterans (REST-V)
- Control condition (Active Comparator): Usual resources
  Interventions: Other: Usual resources

INTERVENTIONS:
Behavioral: Resilience Training for Veterans (REST-V) — A 6-week self-help intervention tailored for post-9/11 Veterans offering guidance on cognitive-behavioral self-management coping strategies plus when and how to access recovery support services including mental health treatment. Materials are sent once a week for 6 weeks, and participants can opt to receive weekly reminder text messages or up to 3 brief telephone support calls.
  Arms: Intervention condition
Other: Usual resources — Standard printed resource/treatment information provided in VHA usual care to post-9/11 Veterans. Covers similar domains as the intervention materials and provides information on a variety of VA and community resources for Veterans. Materials are sent once.
  Arms: Control condition

SUMMARY:
It is important to provide support and resources for the many post-9/11 Veterans with mental health symptoms and poor psychosocial functioning who do not engage in psychotherapy. One of the biggest reasons post-9/11 Veterans do not seek treatment is a preference to handle problems on their own. This study examines a self-help intervention that teaches Veterans healthy coping strategies they can use on their own and how to seek out recovery support services such as mental health treatment or whole-person care if they decide to do so in the future. This study will compare the impact of self-help and standard resources at improving mental health and resource utilization. Two hundred Veterans will complete 6 brief assessments across 40 weeks.

DETAILED DESCRIPTION:
Many post-9/11 Veterans experience impaired psychosocial functioning, due in part to high rates of posttraumatic stress disorder (PTSD) and major depressive disorder (MDD). Less than half of post-9/11 Veterans with these conditions seek mental health treatment, with key barriers being a preference to self-manage and lack of time. Veterans also report difficulty navigating the overwhelming array of resources available. To address this gap for post-9/11 Veterans with unmet mental health needs, the investigators developed a self-help intervention to provide skills for healthy self-management as well as curated guidance on recovery support services that address mental health and broader whole-person functional challenges. The investigators will compare the self-help intervention to a control condition of standard printed resource/treatment information as is provided in usual care. The objective of this clinical trial is to evaluate the efficacy of the intervention (vs. control) at improving psychosocial functional impairment, mental health outcomes, and utilization of cognitive-behavioral coping skills and recovery support services. The investigators will also explore use of coping skills and recovery support services as potential mediators of the intervention. A total of 200 Veterans from the Syracuse and Durham VA healthcare system will complete validated measures in 6 assessments over 40 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Veteran age >= 18 years who served on or after September 11, 2001
* Enrolled at Syracuse or Durham VA Healthcare System (had an encounter in primary care or Military 2VA clinic in past 24 months)
* Screen positive for current symptoms of MDD (PHQ-2) or PTSD (PC-PTSD-5)
* Report current functional impairment (PHQ-9 item 10)

Exclusion Criteria:

* Inability to communicate in English
* Visual impairment that precludes reading self-help materials
* Hearing impairment that precludes completing telephone assessments
* Cognitive impairment that precludes providing informed consent
* Serious mental illness (diagnosis of bipolar disorder or schizophrenia spectrum and other psychotic disorders)
* Engaged in psychotherapy/counseling (>= 2 outpatient therapy visits in past 90 days, scheduled outpatient therapy visit in upcoming 30 days that intends to attend, or psychiatric hospitalization in past 90 days)
* Started or had dosage change in psychotropic medication in the past 4 weeks
* At imminent risk of suicide or has active high-risk for suicide flag

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Inventory of Psychosocial Functioning (IPF) | Weeks 0 to 8, 24, and 40
  An 80-item self-report measure of mental-health related psychosocial functional impairment over the past 30 days. The IPF yields domain scores for up to 7 domains (e.g., work, family, self care), with only those domains relevant for the individual being scored, and an overall score. The overall IPF score is an unweighted average of all calculated domain scores, scaled to a range of 0-100. Higher scores indicate greater psychosocial functional impairment (i.e., lower scores = better functioning).

SECONDARY OUTCOMES:
Brief Symptom Inventory-18 (BSI-18) Global Severity Index | Weeks 0 to 8, 24, and 40
  An 18-item self-report measure of general psychological distress over the past 7 days serves as a cross-cutting mental health outcome not specific to any one mental health diagnosis. The Global Severity Index (GSI) uses all three 6-item subscales (depression, anxiety, somatization), with a total raw score range of 0-72. Raw scores can be converted to T-scores using normative data. Higher scores indicate greater distress.
Patient Health Questionnaire-9 (PHQ-9) | Weeks 0 to 8, 24, and 40
  A 9-item self-report measure of depression symptom severity over the past 2 weeks. The total PHQ-9 score is the sum of all 9 items and can range from 0-27. Higher scores indicate greater depression symptom severity.
Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) | Weeks 0 to 8, 24, and 40
  A 20-item self-report measure of PTSD symptom severity over the past month. The total PCL-5 score is the sum of all 20 items and can range from 0-80. Higher scores indicate greater PTSD symptom severity.
Columbia Suicide Severity Rating Scale (C-SSRS) item 2 | Weeks 0 to 8, 24, and 40
  This self-report item assesses suicidal ideation over the past month with yes or no response options. The full C-SSRS used in VHA will be administered, but this outcome focuses specifically on active suicidal ideation.
Frequency of Actions and Thoughts (FATS) | Weeks 0 to 8
  An 12-item self-report measure of frequency of cognitive-behavioral therapy (CBT) skill utilization over the past week. This measure is sensitive to change from CBT self-help. The total FATS score is the sum of all 12 items (from 4 subscales) and can range from 0 to 48. Higher scores indicate greater frequency of CBT skill utilization.
Recovery Support Services Utilization (RSSU) | Weeks 0 to 40
  The investigators will use cumulative measures of utilization of 3 components across the 40-week study: (1) outpatient mental health treatment (a) within VHA and (b) outside VHA, (2) other relevant VHA whole-person health care, and (3) informal resources. See the other pre-specified outcomes with prefix RSSU below for details on measurement of each component.

OTHER OUTCOMES:
RSSU part 1a: VHA Outpatient Mental Health Treatment | Weeks 0 to 40
  Outpatient mental health treatment within the Veterans Health Administration (VHA) will be assessed using electronic health record (EHR) data. The cumulative total count of three care components occurring across the 40-week study period will be used: (1) encounters of outpatient psychotherapy in primary care (Primary Care Mental Health Integration) or specialty mental health care (outpatient behavioral health, PTSD clinic, substance treatment clinic, or OEF/OIF/OND mental health clinic), (2) encounters of medication management visits with psychiatric prescribers, and (3) psychotropic medication fill or refill not tied to a specific medication management visit (e.g., through primary care). Medication fills/refills identified from the EHR will only be counted if the participant also self-reports taking the medication for at least 4 weeks (assessed every 8 weeks).
RSSU part 1b: Non-VHA Outpatient Mental Health Treatment | Weeks 0 to 40
  Mental health treatment outside VHA will be assessed using self-report occurring every 8 weeks. The cumulative total count of three care components occurring across the 40-week study period will be used: (1) encounters of outpatient psychotherapy (e.g., in community clinic or with therapist in the community), (2) encounters of medication management visits with non-VHA psychiatric prescribers, and (3) psychotropic medication fill or refill not tied to a specific medication management visit (e.g., through non-VHA primary care). Medication fills/refills will only be counted if the participant also self-reports taking the medication for at least 4 weeks (assessed every 8 weeks).
RSSU part 2: Other Relevant VHA Whole-Person Health Care | Weeks 0 to 40
  Other relevant VHA whole-person health care will be assessed using EHR data. The cumulative total count of encounters with the following outpatient services/programs will be used: Whole Health (e.g., Whole Health Coaching, Whole Health classes), Complementary and Integrative Health (acupuncture, biofeedback, clinical hypnosis, massage therapy, meditation, guided imagery, tai chi / qigong, yoga), Social work, Case management (e.g., Military 2 VA, Healthcare for Homeless Veterans), Peer support, Vocational rehabilitation, and Veterans Justice Outreach.
RSSU part 3: Informal Resources | Weeks 0 to 40
  Informal resource use or use of self-directed resources or approaches to support mental health and wellness will be measured via self-report every 8 weeks. To reduce recall bias and assessment reactivity while balancing participant burden, a two-pronged approach will be used. First, open-ended prompts will elicit behaviors over the past 8 weeks related to 5 categories (categorized per codebook): Socialization, VA Resources & Benefits, Health & Wellbeing, Self-Help for Mental Health, and Preparation for Mental Health Treatment. Then, participants will report how often they engaged in each behavior over the past week only using the FATS Likert-scale from 0 (not at all) to 4 (every day). Scores across the 5 categories will be summed for a total score for each time period. An average score will be created using the total scores from weeks 8, 16, 24, 32, and 40. For the exploratory mediation analysis, an average score using the total scores from weeks 8, 16, and 24 only will be created.
Client Satisfaction Questionnaire-8 (CSQ-8) | Post-Treatment (Week 8)
  An 8-item self-report measure of treatment satisfaction will be administered to participants in the intervention condition. The total CSQ-8 score is the sum of all 8 items (4 of which are reverse-scored) and can range from 8 to 32. Higher scores indicate greater treatment satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Robyn L. Shepardson, PhD, Principal Investigator — Syracuse VA Medical Center, Syracuse, NY
Locations (2):
- United States (2):
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying all publications resulting from the research may be shared outside VA. A Limited Dataset (LDS) that does not contain any personally identifiable information (PII) will be created and shared pursuant to a completed written Data Use Agreement (DUA) with the PI.
Time Frame: Requests will be considered beginning 6 months after final publication. Data will be shared upon completion of a written request to the PI and within 90 days of a completed Data Use Agreement.
Access Criteria: The Data Use Agreement (DUA) will appropriately limit use of the dataset and prohibit the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.